CLINICAL TRIAL: NCT03423823
Title: An Active-treatment Study of the Efficacy of Ziv-aflibercept in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Ziv-aflibercept Efficacy in Better Regulating AMD
Acronym: ZEBRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kapil Kapoor (Other)
Responsible Party: Sponsor-Investigator, Kapil Kapoor, Principal Investigator, Wagner Macula & Retina Center
Organization: Wagner Macula & Retina Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZA511293
Record Dates: First submitted 2018-01-23; First posted 2018-02-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Wet Macular Degeneration; Wet Age-related Macular Degeneration
Keywords: Neovascularization
MeSH Terms: conditions — Wet Macular Degeneration; Neovascularization, Pathologic | interventions — aflibercept; Ranibizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Drug Arm (Experimental): Receiving 1.25mg of 0.05mL of Ziv-aflibercept intravitreal injection every month
  Interventions: Drug: Ziv-Aflibercept 25 MG/ML [Zaltrap]
- Control Arm (Other): Receiving bevacizumab, ranibizumab, or aflibercept intravitreal injection every 5 to 12 weeks (varied intervals based on individual need for treatment)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ziv-Aflibercept 25 MG/ML [Zaltrap] — Anti-VEGF injection
  Arms: Study Drug Arm
Drug: Ranibizumab — Anti-VEGF standard of care injection
  Other Names: aflibercept; bevacizumab
  Arms: Control Arm

SUMMARY:
This is a randomized, open-label, interventional, controlled study to determine the effects of Zaltrap on Neovascularized Wet Macular Degeneration as compared to the control anti-vascular endothelial growth factor ("anti-VEGF") injections (bevacizumab, ranibizumab, or aflibercept).

ELIGIBILITY:
Inclusion Criteria:

* Are age 50-99
* Have neovascular Age-related Macular Degeneration ("AMD") with an eye undergoing maintenance treatment with one or more of the following anti-VEGF drugs: bevacizumab, ranibizumab, or aflibercept.
* Have an eye undergoing treatment that is of low visual potential (20/200 Snellen equivalent or worse) and the contralateral eye must have better visual potential.
* Are willing and able to provide signed informed consent and willing to undertake all scheduled study-related assessments, visits, and treatments.
* Have received an intravitreal injection of one of the drugs listed above within 120 days of Day 1 of the trial.
* Both males and females will be enrolled.

Exclusion Criteria:

* Active intraocular inflammation or infection
* History of vitreous hemorrhage within three months prior to Day 1 of the study
* Uncontrolled ocular hypertension or glaucoma in the study eye (defined as Intraocular Pressure ("IOP") >25 mm Hg or a Cup to Disc ratio > 0.8 despite treatment with anti-glaucoma medication) or any such condition which the investigator feels may warrant a glaucoma filtering surgery during the study
* History of stroke within the last three months prior to Day 1 of the study
* History of myocardial infarction within the last three months prior to Day 1 of the study
* Undergone intraocular surgery or laser treatments within the last three months,
* Significant Epiretinal Membrane ("ERM") or Vitreomacular Traction ("VMT") causing distortion of macular anatomy
* No use of ocular corticosteroids within the last six months and no use of systemic corticosteroids at a dose of >10 mg/day
* Not have active malignancies within the last 12 months except appropriately treated carcinoma in situ of the cervix, melanoma, and prostate cancers treated with a curative intent
* Inability to comply with study or follow-up procedures
* Women who may become pregnant or lactating or intend to become pregnant during the study
* Women who are of childbearing potential, including women who have had tubal ligation, must have a blood test within 21 days prior to Day 1 of the study. A woman is considered to not be of childbearing potential if she is postmenopausal or has undergone hysterectomy and/or bilateral oophorectomy. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Efficacy of study drug measured by change in best corrected visual acuity | 18 months
  Change in Snellen equivalent letters from baseline to end of study
Efficacy of study measured by change in central foveal thickness | 18 months
  Change in microns of macular thickness as assessed by Optical Coherence Tomography ("OCT") from baseline to end of study

SECONDARY OUTCOMES:
Safety of study drug as measured by number of adverse events related to study drug | 2.5 years
  adverse events, serious adverse events reported causal to drug

CONTACTS AND LOCATIONS:
Locations (1):
- Wagner Macula & Retina Center, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: No